CLINICAL TRIAL: NCT04391647
Title: Developing Methods to Investigate Additional Opportunities of HPV Vaccination, Including Control of Infection and Transmission, by Using a Cervicovaginal Human Sample, Collected by Urination (HPV-VACPLUS)
Brief Title: Developing Methods to Investigate Additional Opportunities of HPV Vaccination by Using First-void Urine Samples
Acronym: HPV-VACPLUS
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, Professor Pierre Van Damme, MD, PhD, Universiteit Antwerpen
Other Study IDs: B3002020000025
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Human Papilloma Virus Infection
Keywords: First-void urine; Self-sampling; Vaccination; Infectious virions; Neutralizing antibodies; HPV
MeSH Terms: conditions — Papillomavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — First-void urine samples and Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HPV vaccinated group: Women (18-25 years old) whom are previously fully vaccinated with the bivalent (Cervarix), quadrivalent (Gardasil) or nonavalent (Gardasil) prophylactic HPV vaccine.
  No intervention/drug to be administered.
  Interventions: Other: First-void urine collection; Other: Blood draw
- HPV unvaccinated group: Women (18-25 years old) whom are not previously vaccinated with the bivalent (Cervarix), quadrivalent (Gardasil) or nonavalent (Gardasil) prophylactic HPV vaccine.
  No intervention/drug to be administered.
  Interventions: Other: First-void urine collection; Other: Blood draw

INTERVENTIONS:
Other: First-void urine collection — * One time collection of ca. 20 ml of first-void urine with the Colli-PeeTM device (Novosanis) during visit at the Centre for the Evaluation of Vaccination.
  * IF HPV positive and the woman gave consent to be contacted again: Collection of ca. 20 ml of first-void urine with the Colli-PeeTM device (Novosanis) each day during 14 days (n = 14)
  Other Names: FV urine
Other: Blood draw — - One time blood sample collection (5-10 cc) by a study nurse of Centre for the Evaluation of Vaccination.

SUMMARY:
The main objective of this study is to develop protocols using FV urine that investigate in vitro whether infectious virions can be neutralized by HPV vaccination.

DETAILED DESCRIPTION:
In total 50 women will be included in this trial whereof 25 fully vaccinated with a prophylactic HPV vaccine and 25 not vaccinated with a prophylactic HPV vaccine. These women will be asked to collect a first-void urine sample with the Colli-PeeTM device (Novosanis). Hereafter, a blood sample of 5-10 cc will be collected. HPV DNA positive women who gave their consent to be contacted with the results, will later be contacted again and asked to provide additional FV urine samples every day during 2 weeks. For this, urine collection devices (Colli-PeeTM, Novosanis) will be provided by postal mail. The collected urine samples (and blood sample as control for HPV antibodies) will be used for the development of protocols within this project.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-25 years of age
* Sexually active or has been sexually active in the past
* Cases (n=25): fully vaccinated women, i.e. receiving all necessary doses of the HPV vaccine (according to the KCE recommendations) able to prove their vaccination (brand and schedule) with an official document.
* Control group (n=25): women self-reported to be not previously vaccinated with a single dose of any prophylactic HPV vaccine available.
* Willing to give informed consent to the CEV research team.
* Giving consent to the research team (CEV) to contact his/her general practioner and/or gynaecologist to access details of the participants HPV vaccination (schedule) and results of cervical smears/cytology, HPV tests, colposcopy, and biopsy (included in ICF)

Exclusion Criteria:

* Women participating in another clinical study at the same time of this study.
* Women that underwent hysterectomy or were treated for cervical (pre)cancer lesions within the previous six months prior to study enrolment.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In total 50 women will be included in this trial. During their study visit, participants are asked to collect a first-void urine sample with the Colli-PeeTM device. Hereafter, a blood sample of 5-10 cc is collected. Following sample collection, women are asked to fill in a questionnaire. HPV positive women who gave their consent to be contacted with the results will later be again contacted and asked to provide additional FV urine samples every day during 2 weeks.
  Since this is a unique pilot study, no specific data exist for sample size calculation. However, the sample size is estimated based on HPV prevalence results from a surveillance study in Belgium. From the 50 participating women (age 18-25), we expect 20% to be HPV DNA positive.Taking possible dropouts into account, this will lead to approximately 5 HPV infected women to provide samples during 14 days. Ultimately, we will obtain 120 samples to be used to develop the intended protocols.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Protocols to investigate the neutralizing ability of HPV vaccine-induced antibodies | Within 2 years after study completion
  To develop protocols that investigate whether infectious HPV virions may be neutralized by HPV vaccine-induced antibodies, preventing autoinoculation and transmission to sexual partners.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Prof, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universiteit Antwerpen, Antwerp, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: No